CLINICAL TRIAL: NCT04476511
Title: Controlled Randomized Open Label Clinical Study to Compare the Efficacy and the Safety of the Loading Dose Schedules of Vitamin D3 (Colecalciferol) 30,000 IU Product in Deficient Patients
Brief Title: The Efficacy and the Safety of Vitamin D3 30,000 IU for Loading Dose Schedules
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: Pharma Patent Kft. (Unknown)
Responsible Party: Principal Investigator, Istvan Takacs, M.D., DSc., Director of Department, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAT17-LOADS; 2018-000508-40 (EudraCT Number)
Record Dates: First submitted 2019-05-05; First posted 2020-07-20 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D deficiency; vitamin D loading dose
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slower Loading Dose (Active Comparator): 30.000IU cholecalciferol once weekly for ten weeks
  Interventions: Drug: Cholecalciferol
- Moderate Loading Dose (Active Comparator): 30.000IU cholecalciferol twice weekly for five weeks
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — tablet containing 30.000IU cholecalciferol

SUMMARY:
Treatment: A: Slower Loading Group (SLD): 30.000 IU cholecalciferol once weekly for ten weeks, followed by 30.000 IU cholecalciferol every two weeks for four weeks.

B: Moderate Loading Dose group (MLD): 30.000 IU cholecalciferol twice weekly for five weeks, followed by 30.000 IU cholecalciferol every two weeks for four weeks.

Every patients will receive calcium-citrate supplementation if average daily calcium intake does not reach the recommended daily amount.

Setting: two-arms, controlled, randomised, comparative open-label, multicentric clinical trial aimed to assess the comparative efficacy on 25(OH)D elevation and on safety of the two loading dose schedules of 30.000 IU Vitamin D3 oral tablets (administered as "Moderate Loading Dose"or "Slower Loading Dose") combined with an follow-up maintenance period of biweekly administration. The comparative assessment is based on the elevation of 25(OH)D levels due to treatment efficacy from baseline and by the end of the maintenance (biweekly 30.000 IU) period for each treatment groups, and also the ratio of patients in target range (30-50 ng/ml) in order to evaluate the most beneficial "loading dose" schedule. Upon the serum 25(OH)D levels are exceeded the 55ng/ml limits by the end of the loading period the trial subjects should continue with the standard maintenance dose of vitamin D3 for the remaining four weeks of the study. The evaluation of the comparative safety will be done also by controlling the serum and the urinary calcium levels and the registration of adverse drug reaction.

The primary objective is to assess the efficacy of the orally administered loading dose schedules of vitamin D3 in deficient patients. Efficacy is measured as the elevation of 25(OH)D levels compared to baseline.

Rationale: Oral vitamin D3 is the treatment of choice in vitamin D deficiency. The UK NOS guideline recommended where rapid correction of vitamin D deficiency is required, such as in patients with symptomatic disease or about to start treatment with a potent antiresorptive agent, the recommended treatment regimen is based on fixed loading doses followed by regular maintenance therapy. The loading dose regimen to provide a total of approximately 300,000 IU vitamin D, given either as separate weekly or daily doses over 6 to 10 weeks followed by a maintenance therapy comprising vitamin D in doses equivalent to 800-2000 IU daily in general or up to 4,000 IU daily), given either daily or intermittently at higher doses. (NOS guidelines 2014). Recent research on vitamin D and the widening range of therapeutic applications available for cholecalciferol, which can be classified as both a vitamin and a pro-hormone. Additionally, it was now realized that the Food and Nutrition Board's previously defined Upper Limit (UL) for safe intake at 2,000 IU/day was set far too low and that the physiologic requirement for vitamin D in adults may be as high as 5,000 IU/day, which is less than half of the >10,000 IU that can be produced endogenously with full-body sun exposure.

In a recent study showed that the safety of doses over 2000 IU/day-4000 IU/day for 3 months resulting in a ~360,000 UI cumulative dose. According to the study results, for the majority of the patients the 4000 IU/day (360,000 UI cumulative dose) was needed to achieve a 25(OH)D serum concentration above 75nmol/L (30 ng/mL), which is otherwise set as the target value by Endocrine Society Clinical Practice Guideline (Holick 2011b).

Another study (Verussio et al 2014) cited shows the safety and efficacy of 50.000 IU/week for 8 weeks (400,000 UI cumulative dose for 8 weeks), followed by 25,000 IU twice a month which was more effective in raising the 25(OH)D level to the target range (of >30 ng/L) than 25,000 IU twice a month (50,000 IU/ month). In the latter group only 40% of the patients reached the target 25(OH)D levels at 6 months, compared to the 72% in the first group. The study supports efficacy of dosing and safety of the treatment of vitamin D deficiency a 50,000 IU /week loading dose scheme with a 8 weeks cumulative dose of >400,000 UI.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* 25OHD level is no more than 16 ng/ml
* Postmenopausal state or adequate contraception in female patients
* Willing and able to give legal informed consent for study entry

Exclusion Criteria:

* Severe endocrine or metabolic disease, significant metabolic bone disease (except primary age-related osteoporosis)
* significant obesity (BMI >36 kg/m2)
* hypercalcemia at screening or within one year (seCa > 2.60 mmol/l)
* long standing hypercalciuria, kidney stones within 2 years
* sever kidney injury (KDIGO CKD 3 or more)
* chronic disease which significantly affects bone metabolism, vitamin D metabolism or calcium absorption
* significant malabsorption that affects calcium metabolism
* heart failure or angina pectoris
* alcohol or drug abuse
* daily vitamin D intake is more than 1000 IU within 2 months
* suspected or proved pregnancy
* any other symptoms or findings which may interact with the safety of the study drug, evaluated by investigator
* participating in other clinical trial within 3 months of study entry
* planned journey to geographic location with high natural UV-B exposition for mor than 4 days during the study or regular (more than 2 times per month) artificial UV-B exposition (eg. sun parlor)
* Taking prohibited medication:
* glycosides
* magnesium containing medications (eg. antacids)
* cholestyramine and other ion exchange resins, orlistat
* thiazide type diuretics
* microsomal enzyme inductors (eg. anticonvulsants, sedatives)
* corticosteroids
* phosphates
* laxatives
* medications decreasing lipid absorption

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Serum 25-hydroxyvitamin-D increase after loading period | 5/10 weeks
  Serum 25OHD level will be measured at screening, after loading period and after maintenance period

SECONDARY OUTCOMES:
Proportion of subjects reaching target range of serum 25-hydroxyvitamin-D after loading dose | 5/10 weeks
  Serum 25OHD level will be measured at screening, after loading period and after maintenance period. Target range: 30-50 ng/ml
Proportion of subjects remaining in target range of serum 25-hydroxyvitamin-D after maintenance dose | 4 weeks
  Serum 25OHD level will be measured at screening, after loading period and after maintenance period. Target range: 30-50 ng/ml
Efficacy of maintenance dose | 4 weeks
  Serum 25OHD level will be measured at screening, after loading period and after maintenance period. Target range: 30-50 ng/ml
Frequency of adverse events | up to 20 weeks, continuously
  Adverse event recording will be performed at every study visits and unscheduled visits if applicable.
Serum calcium level | up to 20 weeks, continuously
  Serum calcium level will be measured at screening, after loading period and after maintenance period and whenever clinically relevant.
Urinary calcium excretion | whole study
  Urinary calcium level will be measured at screening, after loading period and after maintenance period and whenever clinically relevant from 24 hours collected urine.
Bone turnover markers | up to 20 weeks, continuously
  osteocalcin; collagen-ß-crosslaps

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Takacs, MD, PhD, DSc, Principal Investigator — Semmelweis University
Locations (7):
- Hungary (7):
  - Semmelweis University - Dept. of Medicine and Oncology, Budapest
  - Uno Medical Trials Kft., Budapest
  - Central Hospital of the Hungarian Homeland Defence Forces, Budapest
  - Szalay János Outpatient Clinic, Hajdúnánás
  - Somogy County Kaposi Mór Teaching Hospital, Kaposvár
  - Jutrix Healthcare Ltd., Kecskemét
  - Rub-Int Health Center, Székesfehérvár

IPD SHARING:
Plan to Share IPD: Undecided